CLINICAL TRIAL: NCT05155605
Title: The PATHFINDER 2 Study: Evaluating the Safety and Performance of the GRAIL Multi-Cancer Early Detection Test in an Eligible Screening Population
Brief Title: PATHFINDER 2: a Multi-Cancer Early Detection Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GRAIL, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GRAIL-012
Record Dates: First submitted 2021-11-16; First posted 2021-12-13 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Early Detection of Cancer; Cancer
Keywords: multi-cancer early detection; cancer screening; circulating cell-free tumor DNA; MCED
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Participants 50 years of age or older (Experimental): The study will aim to enroll a diverse participant population generally representative of the US population with respect to race, ethnicity, and sex. The target age categories of 60-69 years and 70-79 years will be enriched to increase the number of cancer events that are observed during the study.
  Interventions: Device: Multi-Cancer Early Detection Test

INTERVENTIONS:
Device: Multi-Cancer Early Detection Test — Blood collection and multi-cancer early detection testing with return of results.

SUMMARY:
This is a prospective, multi-center interventional study of the GRAIL multi-cancer early detection (MCED) test with return of test results for participants enrolled through healthcare systems in North America. The purpose of this study is to evaluate the safety and performance of the GRAIL MCED test in a population of individuals who are eligible for guideline-recommended cancer screening. In cases with a "cancer signal detected" test result, participants will undergo diagnostic procedures based on the test returned cancer signal origin(s) to determine if they have cancer. The number and types of diagnostic procedures required to achieve diagnostic resolution will be assessed. Participant-reported outcomes will be collected at several time points to assess participants' perceptions about the multi-cancer early detection test.

The study will enroll approximately 35,000 and no more than 38,500 participants as defined by eligibility criteria over an anticipated enrollment period of approximately 36 months at up to 40 clinical institutions within North America. Participants will be actively followed for approximately 3 years from the date of their enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be at least 50 years of age, inclusive, at the time of signing the Informed Consent Form (ICF).
2. Participants must be capable of giving signed and legally effective informed consent

Exclusion Criteria:

1. Undergoing or referred for diagnostic evaluation due to clinical suspicion for cancer (e.g., referred to a medical or surgical oncologist, or scheduled for biopsy on the basis of a suspicious imaging abnormality).
2. Personal history of invasive solid tumor or hematologic malignancy, diagnosed within the 3 years prior to expected enrollment date, or diagnosed greater than 3 years prior to expected enrollment date and never treated.

   * Individuals with a diagnosis of non-metastatic basal cell carcinoma and squamous cell carcinoma of the skin are not excluded.
3. Prior/Concurrent Concomitant Therapy (Medications/Treatments):

   * Definitive treatment for invasive solid tumor or hematologic malignancy within the 3 years prior to expected enrollment date. Adjuvant hormone therapy for cancer (e.g. for breast or prostate cancer) is not an exclusion criterion.
4. Individuals who will not be able to comply with the protocol procedures.
5. Individuals who are not currently registered patients at a participating center.
6. Previous or current participation in another GRAIL-sponsored study. "Participation" is defined as having signed consent and provided a blood sample.
7. Previous or current employees or contractors of GRAIL.
8. Current pregnancy (by self-report of pregnancy status)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35885 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Number and type of invasive procedures performed in participants with a cancer signal detected by the multi-cancer early detection (MCED) test and no cancer diagnosis at the time of diagnostic resolution (i.e., false positive test result). | Up to 3 Years
Test performance: diagnosis of invasive cancer, assessed by positive predictive value (PPV). | Up to 3 Years
Test performance: diagnosis of invasive cancer, assessed by negative predictive value (NPV). | Up to 3 Years
Test performance: diagnosis of invasive cancer, assessed by sensitivity. | Up to 3 Years
Test performance: diagnosis of invasive cancer, assessed by specificity. | Up to 3 Years
Test performance: diagnosis of invasive cancer, assessed by cancer signal origin (CSO) accuracy. | Up to 3 Years
Test performance: diagnosis of invasive cancer, assessed by observed cancer detection rate (CDR). | Up to 3 Years
Test performance: diagnosis of invasive cancer, assessed by number needed to screen to detect an invasive cancer (NNS). | Up to 3 Years

SECONDARY OUTCOMES:
Participant-reported anxiety resulting from use of the multi-cancer early detection (MCED) test assessed via questionnaire at various time points during the study. | Up to 3 Years
Participant-reported intention to follow and use guideline recommended cancer screening procedures after use of the multi-cancer early detection (MCED) test assessed via questionnaire at various time points during the study. | Up to 3 Years
Cancer detection rate of confirmatory PET-CT in participants for whom cancer signal origin directed workups do not result in diagnosis of cancer. | Up to 3 Years
Number and type of diagnostic evaluations (imaging procedures, invasive procedures, laboratory test) by predicted cancer signal origin and outcome of diagnostic resolution. | Up to 3 Years
Per-participant radiation exposure during diagnostic evaluation for test positive participants. | Up to 3 Years
Accuracy of initial multi-cancer early detection (MCED) test result and cancer signal origin prediction, among the subset of participants with a research blood draw. | Up to 3 Years
Participants-reported perceptions about the multi-cancer early detection (MCED) test including satisfaction with the MCED tests and attitudes towards subsequent MCED testing assessed via questionnaire at various time points during the study. | Up to 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Celine Marquez, MD, Study Director — GRAIL, Inc.
Locations (56):
- United States (55):
  - Sutter Health, Auburn, California
  - Sutter Health, Davis, California
  - Sutter Health, Elk Grove, California
  - Sutter Health, Fairfield, California
  - HOAG Irvine, Irvine, California
  - HOAG Vivante Newport Mesa, Irvine, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Sutter Health, Modesto, California
  - HOAG Newport Beach, Newport Beach, California
  - Palo Alto Medical Foundation, Palo Alto, California
  - Sutter Health, Sacramento, California
  - PAMF - Santa Cruz, Santa Cruz, California
  - PAMF - Sunnyvale, Sunnyvale, California
  - Sarah Cannon Research Institute - Englewood Primary Care, Englewood, Colorado
  - Medstar Washington Hospital Center, Northwest, District of Columbia
  - Woodlands Medical Specialists, Pensacola, Florida
  - Morehouse School of Medicine, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Ochsner Grove, Baton Rouge, Louisiana
  - Ochsner Lafayette General, Lafayette, Louisiana
  - Ochsner Health, New Orleans, Louisiana
  - Maryland Oncology Hematology, Annapolis, Maryland
  - Henry Ford Macomb, Clinton, Michigan
  - Henry Ford Medical Center Ford Road, Dearborn, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Henry Ford Medical Center Harbortown, Detroit, Michigan
  - Henry Ford Medical Center Detroit North West, Detroit, Michigan
  - Henry Ford Medical Center Sterling Heights, Sterling Heights, Michigan
  - Mayo Clinic - Cancer Center, Rochester, Minnesota
  - Weill Cornell Medicine, New York, New York
  - Flushing Hospital Medical Center, Queens, New York
  - Jamaica Hospital Medical Center, Queens, New York
  - Sarah Cannon Asheville Family Medicine, Asheville, North Carolina
  - Duke University Health System, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - St. Charles Health System, Bend, Oregon
  - Oregon Health & Science University Bay Area Hospital, Coos Bay, Oregon
  - Oregon Health & Science University Knight Cancer Institute, Portland, Oregon
  - SALEM Health, Salem, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute - The Frist Clinic, Nashville, Tennessee
  - Sarah Cannon, Centennial Internal Medicine Continuity Clinic, Nashville, Tennessee
  - Texas Oncology - West Texas, Amarillo, Texas
  - Sarah Cannon, Austin Diagnostic Clinic, Austin, Texas
  - Kelsey-Seybold Clinic Cypress Woods, Houston, Texas
  - Kelsey-Seybold Clinic Holcombe, Houston, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology - Plano West, Plano, Texas
  - University Texas Health San Antonio - Mays Cancer Center, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Inova, Fairfax, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Northwest Cancer Specialists, Vancouver, Washington
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No